CLINICAL TRIAL: NCT07109869
Title: Safety and Efficacy Study to Assess 600 mg Boric Acid Vaginal Inserts With 7- or 14-Days Treatment of Vulvovaginal Candidiasis (VVC)
Brief Title: Safety and Efficacy of Boric Acid Inserts for Treatment of Vulvovaginal Candidiasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: pH-D Feminine Health LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHD-CLIN-BOR302
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Vulvovaginal Candidiases; Vulvovaginal Candidiasis, Genital; Vulvovaginal Candidiasis (VVC)
Keywords: Vulvovaginal Candidiases; VVC
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — boric acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 14 days 600 mg boric acid inserts (Experimental): All patients will self-administer 600 mg boric acid vaginal inserts once daily for 14 days.
  Interventions: Drug: Boric acid
- 7 days 600 mg boric acid inserts followed by 7 days placebo inserts (Experimental): All patients will self-administer 600 mg boric acid vaginal inserts once daily for first 7 days and placebo vaginal inserts for following 7 days.
  Interventions: Drug: Boric acid; Other: Placebo
- 14 days placebo inserts (Placebo Comparator): All patients will self-administer placebo vaginal inserts once daily for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Boric acid — Boric acid vaginal inserts consisting of 600 mg boric acid drug substance filled into white, opaque hypromellose capsules with no additional excipients included in the formulation. Each vaginal insert is sealed into a clear blister cavity.
  Other Names: Orthoboric acid; Hydrogen orthoborate; Trihydroxidoboron
  Arms: 14 days 600 mg boric acid inserts; 7 days 600 mg boric acid inserts followed by 7 days placebo inserts
Other: Placebo — Placebo vaginal inserts containing anhydrous lactose and 1% magnesium stearate are also manufactured and filled into white, opaque hypromellose capsules. Packaged in clear blisters.
  Arms: 14 days placebo inserts; 7 days 600 mg boric acid inserts followed by 7 days placebo inserts

SUMMARY:
This is a Phase 3 clinical study to evaluate the efficacy, safety, and tolerability of boric acid 600 mg vaginal inserts in patients with VVC.

DETAILED DESCRIPTION:
This clinical study will be a multi-center, randomized, placebo-controlled, double-blinded study with a 3-arm design comparing 600 mg boric acid vaginal inserts dosed for 7 or 14 days to placebo. All patients will self-administer vaginal inserts once daily for 14 days.

During self-administration of the study drug, patients will be instructed to utilize an electronic diary (eDiary) to record their daily symptoms from Screening through Day 28 (Visit 5). The following information will be recorded in the eDiary:

* Study drug administration (including time at which study drug was administered, activity following study drug administration, and whether the bladder was emptied prior to administration);
* Vulvovaginal symptoms;
* Any adverse symptoms or symptoms of concern, illnesses, or physical injuries that occur while participating in the clinical study;
* Contraceptive methods utilized;
* Days of menstrual bleeding, including days of heavy menstrual bleeding (defined as "flooding" or bleeding through ≥1 tampon or sanitary pad in 2 hours or less), start date of menstrual cycle, end date of menstrual cycle, and daily quantity of menstrual hygiene product(s) utilized for each day of menses;
* Position (eg, laying down supine, prone, on side) following study drug administration;
* Vulvovaginal sexual activity, including if the sexual activity occurred before or after study drug administration; and
* The presence of any non-exclusionary intravaginal foreign objects (ie, contraceptive vaginal ring, diaphragm, cervical cap, condom, sex toys).

Patients will complete a total of 4 in-person visits at Screening, on Day 7 (Visit 2) (±2 days), Day 15 (Visit 3) (+2 days), and Day 28 (Visit 5) (±2 days), as well as a telephone Follow-Up Visit on Day 21 (Visit 4) (±2 days) (if clinically indicated, the Follow-Up Visit may be performed in-person).

Clinical, mycological, and overall outcomes will be assessed at Day 15 (Visit 3) and Day 28 (Visit 5) for all study arms. If persistent symptoms are present at any visit, a full microbiologic evaluation to assess for persistence of VVC (including KOH wet mount, saline wet mount, and vaginal fungal culture) will be performed. Additionally, screening tests required to rule out other potential causes of symptoms may be performed or repeated at PI or qualified designee discretion. Patients may also be provided with a rescue treatment at PI or qualified designee discretion.

Individual patient participation is expected to be 28 days.

ELIGIBILITY:
Inclusion Criteria

1. Patients who are postmenarcheal, nonpregnant biological females, 12 years of age and older, at Screening;
2. Patients with acute symptomatic VVC infection at Screening, defined as meeting all of the following criteria:

   * A potassium hydroxide (KOH) wet mount or saline wet mount preparation performed from the inflamed vaginal mucosa or secretions demonstrating yeast forms (hyphae or pseudohyphae) of or budding yeast;
   * Vaginal pH ≤4.5; and
   * Total Vulvar Signs and Symptoms (VSS) Scale score of ≥4: vulvovaginal signs (edema, erythema, and excoriation/fissures) and symptoms (vulvovaginal burning, itching, and irritation) as rated using the VSS Scale.
3. Patients aged 21 and older must have cervical cancer screening results meeting the following criteria for inclusion at Screening or within the 1 year prior to Screening: negative for intraepithelial lesion or malignancy or clinically insignificant findings not requiring any further surveillance or treatment beyond a repeat cervical cytology test;

   * Patients between 21 and 29 years of age must have a cervical cancer screening test (Papanicolaou [Pap] smear) performed at Screening or have a documented Pap smear result within 1 year of Screening which must be available for the assessment by the PI or qualified designee at the Screening Visit; and
   * Patients 30 years of age and older must have documented cervical cancer screening tests (Pap smear and high-risk human papillomavirus [HPV]) performed at Screening or have documented results within 1 year of Screening which must be available for the assessment by the PI or qualified designee at the Screening Visit.
4. Patients must be suitable candidates for vaginal treatment, able to insert the study drug, and are comfortable undergoing pelvic exams;
5. Patients willing and able to provide written informed consent or assent (for those 12 to 17 years of age);
6. Patients willing and able to comply with Protocol requirements, instructions, and Protocol-stated restrictions, as determined by the PI;
7. Patients willing and able to give authorization for use of protected health information;
8. Patients of childbearing potential (as defined in Inclusion Criterion 1) must use 1 of the following contraceptive options described below through Day 28 (Visit 5):

   * Copper intrauterine device used continuously and successfully for at least 90 days prior to the first dose of study drug;
   * Levonorgestrel-releasing intrauterine system used successfully for at least 90 days prior to the first dose of study drug;
   * Progestin implant used successfully for at least 90 days prior to the first dose of study drug;
   * Monogamy with a vasectomized male partner (medical assessment of the surgical success of the vasectomy must have occurred at least 6 months prior to the first dose of study drug);
   * Abstinence; or
   * Use of 1 of the following hormonal methods in combination with 1 of the following barrier methods:

     * Hormonal methods
     * Barrier methods
9. Patients must be willing to avoid tampon or menstrual cup use during the Treatment Period (ie, Day 1 to Day 14); and
10. Patients must be willing to abstain from receiving oral intercourse during the Treatment Period (ie, Day 1 to Day 14).

Exclusion Criteria:

1. Patients with known or suspected other active infectious causes of cervicitis, vaginitis, or vulvitis (eg, BV, Chlamydia trachomatis, Neisseria gonorrhoeae, T. vaginalis, or genital lesions consistent with HPV, herpes simplex, syphilis, chancroid, etc) based on the results of clinical assessments, in-clinic microscopic assessments (eg, clue cells or trichomonads detected on saline wet mount), and/or rapid diagnostic tests (RDTs) performed prior to enrollment (eg, OSOM® test, etc);
2. Patients who have undergone any vaginal rejuvenation procedure (ie, laser) within 4 weeks prior to Screening or plan to undergo a vaginal rejuvenation procedure prior to completion of the last planned assessment;
3. Patients who will undergo evaluation or treatment during the clinical study for abnormal cytology or findings from high-risk HPV testing or Pap test finding;
4. Patients diagnosed with BV, determined by meeting 3 of the 4 Amsel's criteria:

   * A fishy odor of the vaginal discharge before or after the addition of a drop of 10% KOH (ie, a positive whiff test);
   * Homogenous, thin discharge (milk-like consistency) that smoothly coats the vaginal walls;
   * At least 20% of epithelial cells are clue cells (eg, vaginal epithelial cells studded with adherent bacteria) on saline wet mount microscopic evaluation of vaginal discharge; or
   * pH of vaginal fluid >4.5.
5. Patients currently undergoing treatment for or with a history of treatment for cervical, vaginal, or vulvar cancer;
6. Patients using any systemic (eg, oral or injectable) corticosteroid treatment during the study or within 30 days prior to Screening;
7. Patients using topical steroids applied to the vulvar or vaginal regions during the study or within 7 days prior to Screening;
8. Patients using any systemic (eg, oral or injectable) or topical (applied to the vulvar or vaginal regions) antimicrobials including antifungal, antiviral, antibacterial, or anti-trichomonal drugs during the clinical study or within 14 days prior to Screening;
9. Patients using any prescription (eg, vaginal estrogen, ospemifene, prasterone) or non-prescription intravaginal or vulvar product (eg, vitamin E gel capsules [vaginal inserts], lubricants, moisturizers, douches, creams, or spermicides) within 7 days prior to Screening and through Day 28 (Visit 5);
10. Patients unwilling to refrain from the use of intravaginal products (eg, douches, creams, spermicides, yoni eggs, tampons, menstrual cups, and any other such intravaginal product that, in the opinion of the PI, would be considered exclusionary) during the Treatment Period, inclusive of Day 14;
11. Patients with a current immunocompromising condition (ie, HIV, end-stage renal disease);
12. Patients using any immunosuppressive medication (included, but not limited to, carbamazepine, cyclosporine, tacrolimus, methotrexate, 6 mercaptopurine, or mycophenolate) or radiation treatment within 3 months prior to Screening or during the clinical study;
13. Patients with a history of pelvic radiation treatment;
14. Patients with a clinically significant major organ disease, cancer, infection (except acute VVC), or other condition that may affect the clinical assessment of VVC or render the patient a poor study candidate, per the PI's judgment;
15. Patients with any comorbid condition that would preclude the safe participation of the patient in the clinical study or would prevent the patient from meeting the clinical study requirements, per the PI's judgment;
16. Patients with diabetes mellitus type I, use of insulin (current or anticipated need during the study), or poorly-controlled diabetes mellitus type II, defined as (hemoglobin A1c [(HbA1c]) of 10% or higher result within the prior 6 months) or at Screening;
17. Patients with any laboratory abnormality that, in the opinion of the PI, would likely introduce additional risk to the patient or might interfere with data interpretation. The findings noted below are particularly exclusionary:

    * Serum alanine aminotransferase ≥2.5 × the upper limit of normal (ULN) of the reference range;
    * Serum aspartate aminotransferase ≥2.5 × the ULN of the reference range; or
    * Serum total bilirubin ≥2 × the ULN of the reference range, unless the elevation is consistent with Gilbert's syndrome
18. Patients with a known history of HIV, hepatitis B, or hepatitis C virus (HCV), or a positive test for HIV antibody, hepatitis B surface antigen, or HCV antibody;
19. Patients who are pregnant (ie, a positive pregnancy test at Screening), lactating, or planning to become pregnant during the clinical study period;
20. Patients with a planned surgery or other medical procedure that would impact compliance with the Protocol, per the PI's discretion;
21. Patients with a current or recent history (eg, the past 12 months) of substance abuse (including alcohol) or any other medical, psychiatric, or other condition that, in the PI's opinion, would preclude compliance with the Protocol;
22. Patients currently participating or had participated in another clinical study within the 30 days prior to Screening;
23. Patients currently have or expect, within the Treatment Period, to have heavy menstrual bleeding (defined as "flooding" or bleeding through ≥1 tampon or sanitary pad in 2 hours or less with most periods) or a menstrual duration >7 days; or
24. Patients currently have or suspect to have an active urinary tract infection (UTI) based on urinalysis and clinical assessment.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Patients who are postmenarcheal, nonpregnant biological females
Enrollment: 201 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with the absence of all signs and symptoms of vulvovaginal candidiasis | 28 days (+ 2 days)
  The proportion of patients who achieve clinical cure (defined as the absence of all signs and symptoms of vulvovaginal candidiasis (VVC) [ie, composite VSS score = 0] in the absence of additional antifungal treatment), at the test-of-cure (TOC) visit. This is the proportion of patients in the modified ITT (mITT) Population with clinical cure.
  * Signs: vulvovaginal edema, erythema, excoriation/fissures;
  * Symptoms: vulvovaginal itching, burning, irritation; and
  * Severity of each sign and symptom graded on a 0 to 3 rating scale:
    * Absent = 0;
    * Mild = 1;
    * Moderate = 2; or
    * Severe = 3.

SECONDARY OUTCOMES:
Proportion of patients with clinical cure at the end-of-treatment visit | 15 days (+ 2 days)
  Proportion of patients with clinical cure at the end-of-treatment visit in the modified intent to treat (mITT) and clinically evaluable (CE) populations.
Proportion of patients with clinical cure at the test-of-cure visit | 28 days (+ 2 days)
  Proportion of patients with clinical cure at the test-of-cure (TOC) visit in the per protocol and clinically evaluable (CE) populations.
Proportion of patients with mycological eradication at the end-of-treatment visit | 14 days (+ 2 days)
  Proportion of patients with mycological eradication at the end-of-treatment (EOT) visit in the modified intent to treat (mITT) population.
Proportion of patients with mycological eradication at the test-of-cure visit | 28 days (+ 2 days)
  Proportion of patients with mycological eradication at the test-of-cure (TOC) visit in the modified intent to treat (mITT) and clinically evaluable (CE) populations.
Proportion of patients with overall cure at the end-of-treatment visit | 15 days (+ 2 days)
  Proportion of patients with both clinical cure and mycological eradication (ie, overall cure) at the end-of-treatment (EOT) visit in the modified intent to treat (mITT) and clinically evaluable (CE) populations.
Proportion of patients with overall cure at the test-of-cure visit | 28 days (+ 2 days)
  Proportion of patients with both clinical cure and mycological eradication (ie, overall cure) at the test-of-cure (TOC) visit in the modified intent to treat (mITT) and clinically evaluable (CE) populations.
Proportion of patients with clinical cure at both the end-of-treatment and test-of-cure visits | 28 days (+ 2 days)
  Proportion of patients with clinical cure at both the end-of-treatment (EOT) and test-of-cure (TOC) visits in the modified intent to treat (mITT) and clinically evaluable (CE) populations.
Proportion of patients with composite vulvovaginal signs and symptoms score >0 but <4 in the absence of additional antifungal treatment at the end-of-treatment visit | 15 days (+ 2 days)
  Proportion of patients with composite vulvovaginal signs and symptoms (VSS) score >0 but <4 in the absence of additional antifungal treatment at the end-of-treatment (EOT) visit in the modified intent to treat (mITT) population.
  The VSS scale is a standardized, predefined scale for which each sign and symptom is given a numerical rating based on severity (absent = 0; mild = 1; moderate = 2; and severe = 3) to calculate a total composite VSS score (range of 0 to 18). Signs include edema, erythema, and excoriation/fissures. Symptoms include vulvovaginal burning, itching, and irritation.
Proportion of patients with composite vulvovaginal signs and symptoms score >0 but <4 in the absence of additional antifungal treatment at the test-of-cure visit | 28 days (+ 2 days)
  Proportion of patients with composite vulvovaginal signs and symptoms (VSS) score >0 but <4 in the absence of additional antifungal treatment at the test-of-cure (TOC) visit in the modified intent to treat (mITT) and clinically evaluable (CE) populations.
  The VSS scale is a standardized, predefined scale for which each sign and symptom is given a numerical rating based on severity (absent = 0; mild = 1; moderate = 2; and severe = 3) to calculate a total composite VSS score (range of 0 to 18). Signs include edema, erythema, and excoriation/fissures. Symptoms include vulvovaginal burning, itching, and irritation.
Proportion of patients with individual signs and symptoms scores that remain >0, but have improved from baseline in the absence of additional antifungal treatment | 28 days (+ 2 days)
  Proportion of patients with individual signs and symptoms scores that remain >0, but have improved from baseline in the absence of additional antifungal treatment, meeting the following criteria in the modified intent to treat (mITT) and clinically evaluable (CE) populations:
  * Baseline mild (severity = 1) rating resulting in an absence rating at the end-of-treatment (EOT) and test-of-cure (TOC) visits;
  * Baseline moderate (severity = 2) rating resulting in a mild (severity = 1) or absence (severity = 0) rating at the EOT and TOC visits; or
  * Baseline severe (severity = 3) rating resulting in a moderate (severity = 2), mild (severity = 1), or absence (severity = 0) rating at the EOT and TOC visits.
Proportion of patients with complicated vulvovaginal candidiasis | 28 days (+ 2 days)
  Proportion of patients with complicated vulvovaginal candidiasis (VVC) not meeting any study exclusion criteria (that is, VVC with the isolation of non-albicans Candida species [eg, Candida glabrata], severe symptoms [ie, vulvovaginal signs and symptoms (VSS) score ≥7 at screening], and/or recurrent episodes [defined as 3 or more episodes of symptomatic infection within 1 year, inclusive of the study-qualifying infection]) with clinical cure, mycological cure, and overall cure at the end-of-treatment (EOT) and test-of-cure (TOC) visits in the modified intent to treat (mITT) and clinically evaluable (CE) populations.
  The VSS scale is a standardized, predefined scale for which each sign and symptom is given a numerical rating based on severity (absent = 0; mild = 1; moderate = 2; and severe = 3) to calculate a total composite VSS score (range of 0 to 18). Signs include edema, erythema, and excoriation/fissures. Symptoms include vulvovaginal burning, itching, and irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Manager, Study Chair — Medpace GmbH
Locations (20):
- United States (20):
  - Alliance for Multispecialty Research - Mobile, Mobile, Alabama
  - Abby's Research Institute, Phoenix, Arizona
  - Century Research Institute, Inc, Huntington Park, California
  - Matrix Clinical Research, Los Angeles, California
  - Project 4 Research Inc, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Felicidad Medical Research, LLC, Miami, Florida
  - Better Life Clinical Research, LLC, Tampa, Florida
  - Helping Hands Health Center, Tampa, Florida
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Clinical Trials Management, LLC - Northshore, Covington, Louisiana
  - Praetorian Pharmaceutical Research, Marrero, Louisiana
  - Revive Research Institute, Inc., Dearborn Heights, Michigan
  - Cross Creek Medical Clinic, PA, Fayetteville, North Carolina
  - Unified Women's Clinical Research - Raleigh, Raleigh, North Carolina
  - Unified Women's Clinical Research - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Nexgen Research, Lima, Ohio
  - Jackson Clinic, Jackson, Tennessee
  - TMC Life Research, Inc, Houston, Texas
  - National Clinical Trials - VA, Reston, Virginia

IPD SHARING:
Plan to Share IPD: Undecided